CLINICAL TRIAL: NCT07159542
Title: MUSic Listening Impact on QUality of Life, Brain and Burnout of ALzheimer' Patients Informal Caregivers
Acronym: MUSIQUAL+
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-0160; 2024-A01480-47 (Registry Identifier: National)
Record Dates: First submitted 2025-08-26; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer Dementia (AD); Caregivers
Keywords: Caregivers; Music intervention; Alzheimer
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CONTROL (Active Comparator): listening podcast (verbal) in dyads during 12 weeks
  Interventions: Behavioral: listening intervention; Behavioral: Neuropsychology assessment; Other: brain imaging examination
- MUSIC (Active Comparator): listening music during 12 weeks caregivers alone
  Interventions: Behavioral: listening intervention; Behavioral: Neuropsychology assessment; Other: brain imaging examination
- MUSIC+ (Experimental): listening music in dyads during 12 weeks
  Interventions: Behavioral: listening intervention; Behavioral: Neuropsychology assessment; Other: brain imaging examination

INTERVENTIONS:
Behavioral: listening intervention — Music or podcast listening intervention
Behavioral: Neuropsychology assessment — Neuropsychology assessment
Other: brain imaging examination — EEG: recording of neural dynamic

SUMMARY:
Although life expectancy is increasing, the risk of dependence and/or loss of autonomy is increasing too with ageing. Alzheimer's disease affects many people and this kind of disease is constantly growing. Today, relatives of these sick people are increasingly taking on the role of carer to help them remain at home as long as possible. This situation of assistance has often a negative impact on the quality of life of the caregiver, which in some cases can lead to the caregiver burnout and increase the risk factors for developing pathological ageing. This situation can also damage the relationship and the quality of interactions between patient/caregiver dyad. Non-pharmacological therapies and the use of digital tools appear to be promising avenues to fight psychological distress and social isolation, but also to improve the quality and duration of homecare services, by promoting the autonomy of the patient. The MUSIQUAL+ study aims to evaluate the impact of music listening offered to caregivers, alone or with their sick relative, on the quality of life and the exhaustion felt by the caregiver. Three times 20-minute sessions a week of music listening at home through the use of a tablet application, for 12 weeks, will be proposed. In addition to the collection of subjective feelings of the caregivers, a neuropsychological evaluation of the patient and the caregiver will be carried out on 90 dyads divided. Finally, in order to better understand the cerebral mechanisms involved and to provide evidence of the effect of this intervention, an EEG recording will be made before and after the musical listening. This study proposes a therapeutic and preventive alternative to drug treatments and to the currently unsatisfactory support of patients and their caregivers in distress; its benefits will be assessed too.

ELIGIBILITY:
Inclusion Criteria:

* Native language: French
* Medical, neurological, neuropsychological and neuroradiological depth in accordance with the criteria for inclusion and exclusion-specific population, that is to say:

  * Informal Caregivers: Being a carer for someone with neurodegenerative cognitive disorders (NCD), living at home, without memory complaints, normal performances compared to the age and the educational level for all tests of the diagnostic battery.
  * Patients with neurodegenerative cognitive disorders: presenting neurodegenerative cognitive disorders, have an identified informal caregiver.

Exclusion Criteria:

* A chronic neurological, psychiatric, endocrine, hepatic or infectious complaint
* A history of major disease (an uncontrolled diabetes, a lung, heart, metabolic, hematologic, endocrine disease or a severe cancer);
* A medication that may interfere with memory or metabolic measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
EEG phase lag index differences between group | through study completion, an average of 12 weeks
  Functional connectivity (EEG phase lag index (PLI) in each frequency band) differences between group

CONTACTS AND LOCATIONS:
Locations (1):
- PFRS Caen France, Caen, France

IPD SHARING:
Plan to Share IPD: No